CLINICAL TRIAL: NCT00022399
Title: A Randomized, Placebo-Controlled Trial Of Celecoxib In Men Pre-Prostatectomy For Clinically Localized Adenocarcinoma Of The Prostate: Evaluation Of Drug-Specific Biomarker Modulation
Brief Title: Celecoxib Compared With No Treatment Before Surgery in Treating Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: J0007; P50CA058236 (NIH); P30CA006973 (NIH); CDR0000068812; 00-03-08-01 (Other: JHM IRB); NCI-N01-95129; NCI-P01-0186
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Celecoxib (Experimental): Participants receive celecoxib 400mg by mouth twice daily for 4 to 6 weeks prior to standard-of-care prostatectomy.
  Interventions: Drug: celecoxib
- Placebo-control (Placebo Comparator): Participants receive placebo for 4 to 6 weeks prior to standard-of-care prostatectomy.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: celecoxib — 400mg PO twice daily for 4-6 weeks up to 8 hours prior to prostatectomy.
  Other Names: celebrex
  Arms: Celecoxib
Drug: Placebos — Placebo PO twice daily for 4-6 weeks up to 8 hours prior to prostatectomy.
  Arms: Placebo-control

SUMMARY:
RATIONALE: Celecoxib may be an effective treatment for early stage prostate cancer. It is not yet known if celecoxib is more effective than no treatment before surgery for prostate cancer.

PURPOSE: Randomized phase I trial to determine the effectiveness of celecoxib given before surgery to remove the prostate in treating patients who have localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare biomarker modulation (prostaglandin levels) in tissue samples of patients with localized prostate cancer treated with neoadjuvant celecoxib vs placebo followed by prostatectomy.
* Compare the effect of these regimens on angiogenic factors within the prostate in these patients.
* Determine the pharmacokinetic and pharmacodynamic effects of celecoxib in these patients.
* Compare the toxicity profiles of these regimens in these patients.
* Compare the compliance of patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral neoadjuvant celecoxib twice daily.
* Arm II: Patients receive oral neoadjuvant placebo twice daily. Treatment in both arms continues for at least 4 weeks followed by prostatectomy.

Patients are followed within 1 month and then at 3 months.

PROJECTED ACCRUAL: A total of 60-70 patients (at least 30 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed localized adenocarcinoma of the prostate with one or more of the following:

  * Gleason sum at least 7
  * Prostate-specific antigen (PSA) at least 15 ng/mL
  * Clinical stage T2b or T2c (stage II)
  * Any combination of PSA, clinical stage, or Gleason sum with an estimated risk of capsular penetration greater than 45%
* At least 3 positive core biopsies
* Planned radical prostatectomy
* No metastatic disease secondary to prostate cancer

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 9 g/dL
* No history of bleeding disorders

Hepatic:

* Bilirubin less than 1.5 mg/dL
* AST/ALT less than 1.5 times upper limit of normal
* No viral hepatitis

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 50 mL/min

Other:

* No history of hypersensitivity and/or adverse reactions to salicylates
* No allergy to sulfa-containing medications
* No other active malignancy within the past 5 years except superficial bladder cancer or nonmelanoma skin cancer
* No medical or psychiatric problem that would preclude study participation
* No active infection
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunologic therapy for prostate cancer

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* No prior androgen ablation for prostate cancer
* At least 4 weeks since prior hormonal therapy and recovered
* At least 30 days since prior chronic use (more than 3 times per week for more than 2 weeks) of glucocorticoids
* No concurrent glucocorticoids

Radiotherapy:

* At least 4 weeks since prior radiotherapy to the pelvis or surrounding tissues and recovered

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior major surgery and recovered

Other:

* No prior investigational therapy for prostate cancer
* No prior or concurrent chronic anticoagulants
* No prior cyclo-oxygenase-2 inhibitor therapy (e.g., rofecoxib or celecoxib)
* At least 4 weeks since prior initiation of vitamins (except multivitamin) or herbs with known effects on prostate function (PSA)
* At least 30 days since prior chronic use (more than 3 times per week for more than 2 weeks) of aspirin (greater than 100 mg/day) or non-steroidal anti-inflammatory drugs (NSAIDs)
* At least 24 hours since prior use and no concurrent use of any of the following:

  * Over-the-counter (OTC) or prescription products containing aspirin or NSAIDs; OTC products containing bismuth subsalicylate, sodium salicylate, and/or magnesium salicylate; choline salicylate; ranitidine; cimetidine; famotidine; or lansoprazole
* No aspirin (100 mg/day) within 1 week prior to surgery
* No concurrent addition of vitamins or herbal supplements

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2002-04-25; Primary Completion 2005-01-31 (Actual); Study Completion 2005-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Carducci, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Antonarakis ES, Heath EI, Walczak JR, Nelson WG, Fedor H, De Marzo AM, Zahurak ML, Piantadosi S, Dannenberg AJ, Gurganus RT, Baker SD, Parnes HL, DeWeese TL, Partin AW, Carducci MA. Phase II, randomized, placebo-controlled trial of neoadjuvant celecoxib in men with clinically localized prostate cancer: evaluation of drug-specific biomarkers. J Clin Oncol. 2009 Oct 20;27(30):4986-93. doi: 10.1200/JCO.2009.21.9410. Epub 2009 Aug 31. PMID 19720908